CLINICAL TRIAL: NCT05273372
Title: A Randomized Double Blind Placebo Controlled Trial to Determine the Effects of Oxaloacetate on Improving Fatigue in ME/CFS
Brief Title: RESTORE ME -- RCT of Oxaloacetate on Improving Fatigue in ME/CFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terra Biological LLC (Industry)
Collaborators: Bateman Horne Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TB-2022-AEO ME/CFS v1.6
Record Dates: First submitted 2022-02-18; First posted 2022-03-10 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-11

CONDITIONS: Myalgic Encephalomyelitis; Chronic Fatigue Syndrome; Fatigue
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue | interventions — Oxaloacetic Acid

STUDY DESIGN:
Intervention Model Description: Placebo-controlled double blinded 2 arm study. 40 patients in treatment arm, 40 patients in placebo arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 2 sets of bottles will be delivered to the Bateman Horne Center-- Group 1 and Group A. One of the groups will contain the active, the other the placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxaloacetate (Experimental): 500 mg anhydrous enol-oxaloacetate in hypromellose capsules (veggie caps). 2 capsules with breakfast and 2 capsules with lunch (1,000 mg BID) for 90 days.
  Interventions: Other: Medical Food - Anhydrous Enol-Oxaloacetate
- Placebo (Placebo Comparator): 500 mg white rice flour in hypromellose capsules (veggie caps). 2 capsules with breakfast and 2 capsules with lunch (1,000 mg BID) for 90 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Placebo treatment with the food white rice flour. 1,000 mg BID
  Other Names: White Rice Flour
  Arms: Placebo
Other: Medical Food - Anhydrous Enol-Oxaloacetate — Active treatment with oxaloacetate. 1,000 mg BID
  Other Names: Oxaloacetate
  Arms: Oxaloacetate

SUMMARY:
There is no approved treatment for fatigue in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS), a condition with as many as 2.5 million people in the US. Initial case studies have shown an improvement in fatigue in ME/CFS with anhydrous enol-oxaloacetate (AEO).

This randomized, double blinded, placebo controlled trial will seek to further evaluate the efficacy of AEO to reduce fatigue in ME/CFS, based on change in the Chalder Fatigue Score (Likert Scoring) of the AEO group against the placebo group at 90 days.

As secondary evaluations on other core ME/CFS symptoms, the investigators are measuring the health related quality of life as assessed by the SF-36, hours of upright activity, functional capacity (activity, steps, cognition, and heart rate variability), and general health status (global change, vitals)

Finally, this test will gain preliminary insights on the safety, tolerability, and efficacy of AEO in ME/CFS patients.

DETAILED DESCRIPTION:
Anhydrous Enol-Oxaloacetate is a patented thermally stabilized oxaloacetate compound with a multiple year stability rating that when ingested forms bioidentical oxaloacetate. Oxaloacetate is a human metabolite involved in many biochemical reactions in the cytosol and mitochondrial, and is key to energy production.

The investigators will conduct a randomized double blind placebo control trial to determine the effects of AEO on improving fatigue in ME/CFS. The primary measurement with be the Chalder Fatigue Score. The trial will be performed at one site, the Bateman Horne Center, which specializes in the treatment of ME/CFS. The trial will also evaluate the effect of AEO on other core ME/CFS symptoms, health related quality of life as assessed by the SF-36, hours of upright activity, functional capacity (upright activity, steps, cognition, and heart rate variability) and general health status (global change, vitals). The trial will also gain preliminary insights on the safety, tolerability, and efficacy of AEO in ME/CFS patients.

Treatment in the trial will be over a 90-day period for each patient. Participants will be primarily recruited from Bateman Horne's current patients and BHCs databases of research participants. Participants will be screened by telephone for potential eligibility, and if eligible, will be invited to an in person visit at Bateman Horne Center to further confirm eligibility and obtain informed consent. Evaluation will include assessment of vital signs, weight, determination of 5-minute a standard 12-lead electrocardiogram to determine heart rate variability (HRV), cognitive testing, and collection of a fasting blood. Women who could potentially be pregnant will undergo pregnancy testing. Participants will complete baseline questionnaires that assess ME/CFS symptoms, and will undergo cognitive testing, along with a blood draw for biobanking for future banking and eventual metabolomic testing that could include assays such as metabolomics, lipidomics and transcriptomics. Subjects will be provided with a device to wear on their ankle that will determine daily steps and upright activity.

On Visit 1 participants will receive two bottles of 90-day supply of the study capsules treatment and will be instructed to take two 500 mg capsule at breakfast and again at lunch. When participants return for Visit 2, they will bring the bottles of study product with them. BHC will take account of the initial 4-week supplies of the product remaining and provide the participant with another bottle of product. When participants return for study dietary supplement will be distributed at Visit 2 and Visit 3, they will bring the bottles of study project with them, BHC will take account of the remaining product and provide the participant with another bottle. For the final Visit 4, participant will bring the bottles of study product with them and BHC will take account of remaining study product.

Participants will be contacted once every two weeks by the study coordinator to assess for any side effects or difficulty taking the study dietary supplement. They will be asked to return for an in person visit every 4 weeks for 90 days at which time any symptoms or toxicities will be formally documented, and they will complete follow-up questionnaires to assess symptoms, cognition, and heart rate variability. After 12 weeks there will be a final in person visit with a final physical examination, 5-minute HRVEKG, cognitive testing, and symptom assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all of the following criteria are eligible to participate in the study:

  * Provision of signed and dated informed consent form
  * Ability to read, understand or speak English
  * Diagnosed with ME/CFS and meet the IOM Diagnostic Criteria for ME/CFS (2015)
  * Relatively stable state of illness for the past 3 months that is characterized by >2 and <6 hours of daily upright activity
  * Male or female, between the ages of 18 and 65 years old
  * No evidence of active infection with SARS-CoV-2 documented by a negative test at Visit 1
  * Agree to refrain from taking medications that would affect assessment of the effectiveness of study dietary supplement for the duration of the study
  * Females of childbearing potential should be on adequate contraception such as oral, implantable, injectable or transdermal hormonal contraceptives (should have been used for a minimum of one full cycle prior to administration of study drug), intrauterine devices (IUD), vasectomized partner, double barrier method (male or female condom, sponge, diaphragm or vaginal ring with simultaneous use of spermicidal jelly or cream)
  * Each patient of child-bearing potential must have a negative urine pregnancy test at Visit 1. The urine test at Visit 1 must both be confirmed negative prior to randomization. Women of child-bearing potential will have a urine pregnancy test at each visit (2-4) and it must be negative to continue. Women who are confirmed to be of non-childbearing potential do not require pregnancy testing. To be considered of non-child-bearing potential, the patient must be: post-menopausal (defined as no menses for at least one year); or surgically sterile (s/p hysterectomy, bilateral oophorectomy or bilateral tubal ligation at least 6 months prior to randomization); or at least 3 months s/p a non-surgical permanent sterilization procedure
  * History of fatigue and post-exertional malaise (PEM)
  * Stated willingness to comply with all study procedures and remain available for the study duration
  * Have mobile (smart) phone and access to the internet
  * Willingness to wear a device on their ankle

Exclusion Criteria:

* A patient who meets any of the following criteria will be excluded from participation in this study:

  * A positive rapid COVID-19 antigen test at Visit 1
  * Alternate medical or psychiatric illness that could explain the ME/CFS symptoms
  * Severe ME/CFS with less than 2 hours of upright activity a day
  * Active or uncontrolled co-morbidities which in the opinion of the PI may interfere with the ability of the patient to participate in the study. Co-morbidities may include acute infection, Crohn's disease, diabetes mellitus (Type 1 or Type 2, evidenced by a history of HbA1c > 7 at any time), Guillain-Barre syndrome, lupus, multiple sclerosis, myasthenia gravis, rheumatoid arthritis, or other such diseases that may be exclusionary. Particularly conditions or medications that cause immunodeficiency or immunosuppression will be excluded. Examples of such conditions can be found in the tables "Causes of Secondary Immunodeficiency" and "Some Drugs that Cause Immunosuppression" in the "Merck Manual"
  * Body Mass Index > 35
  * Participating in another clinical treatment trial, or symptoms improving as a result of treatment intervention in the past 3 months
  * Current treatment with stimulants including methylphenidate, amphetamine-dextroamphetamine, lisdexamfetamine, modafinil, armodafinil
  * Pregnancy, or while breast feeding. Women should not be enrolled within 6 months of giving birth and within 3 months of cessation of breast feeding.
  * History of:
* Major depression with psychotic or melancholic features before the diagnosis of ME/CFS, or active depression (major depression with psychotic or melancholic features) as determined by self-report
* Untreated endocrine diagnoses including hypothyroidism (Hashimoto's, etc.), Grave's disease, adrenal insufficiency, hypogonadism (testosterone deficiency), diabetes mellitus or insipidus
* Significant head injury in the last 3 years, concussion with loss of consciousness, brain surgery, an automobile accident with head/neck injury, and/or other traumatic brain injury
* A supra-ventricular tachycardia or ventricular tachycardia, e.g., atrial fibrillation or flutter, paroxysmal atrial fibrillation, junctional tachycardia, ventricular tachycardia
* Symptomatic hypotension defined as rested sitting systolic BP < 100 mmHg or rested sitting diastolic BP < 60 mmHg
* Substance abuse in the past 12 months as determined by self-report • Improvement in overall ME/CFS symptoms as a result of any treatment intervention in the past 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Reduction of Fatigue | 90 days
  Reduction in fatigue, Likert Scoring, on the Chalder Fatigue Scale 0-33 Point Scale, with 0 being no fatigue, and 33 being maximum measurable fatigue

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 90 days
  Comparison of adverse events in the treatment group as opposed to the placebo group
Physical Functioning on the SF-36 | 90 days
  Evaluation of the SF-36 for physical functioning, role physical, bodily pain, and others
Patient Global Impression of Change Questionnaire, 7 point scale, -3 to +3, with the higher score indicating more improvement | 90 days
  Measurement of patlient's rating of overall improvement

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne D Vernon, Ph.D., Principal Investigator — Bateman Horne Center
Locations (1):
- Bateman Horne Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided
At this time the IPD is not available to other researchers.

REFERENCES:
- [Background] Germain A, Ruppert D, Levine SM, Hanson MR. Metabolic profiling of a myalgic encephalomyelitis/chronic fatigue syndrome discovery cohort reveals disturbances in fatty acid and lipid metabolism. Mol Biosyst. 2017 Jan 31;13(2):371-379. doi: 10.1039/c6mb00600k. PMID 28059425
- [Background] Germain A, Barupal DK, Levine SM, Hanson MR. Comprehensive Circulatory Metabolomics in ME/CFS Reveals Disrupted Metabolism of Acyl Lipids and Steroids. Metabolites. 2020 Jan 14;10(1):34. doi: 10.3390/metabo10010034. PMID 31947545
- [Background] Committee on the Diagnostic Criteria for Myalgic Encephalomyelitis/Chronic Fatigue Syndrome; Board on the Health of Select Populations; Institute of Medicine. Beyond Myalgic Encephalomyelitis/Chronic Fatigue Syndrome: Redefining an Illness. Washington (DC): National Academies Press (US); 2015 Feb 10. Available from http://www.ncbi.nlm.nih.gov/books/NBK274235/ PMID 25695122
- [Background] Keller BA, Pryor JL, Giloteaux L. Inability of myalgic encephalomyelitis/chronic fatigue syndrome patients to reproduce VO(2)peak indicates functional impairment. J Transl Med. 2014 Apr 23;12:104. doi: 10.1186/1479-5876-12-104. PMID 24755065
- [Background] Mandarano AH, Maya J, Giloteaux L, Peterson DL, Maynard M, Gottschalk CG, Hanson MR. Myalgic encephalomyelitis/chronic fatigue syndrome patients exhibit altered T cell metabolism and cytokine associations. J Clin Invest. 2020 Mar 2;130(3):1491-1505. doi: 10.1172/JCI132185. PMID 31830003
- [Background] McHorney CA, Ware JE Jr, Lu JF, Sherbourne CD. The MOS 36-item Short-Form Health Survey (SF-36): III. Tests of data quality, scaling assumptions, and reliability across diverse patient groups. Med Care. 1994 Jan;32(1):40-66. doi: 10.1097/00005650-199401000-00004. PMID 8277801
- [Background] Nagy-Szakal D, Barupal DK, Lee B, Che X, Williams BL, Kahn EJR, Ukaigwe JE, Bateman L, Klimas NG, Komaroff AL, Levine S, Montoya JG, Peterson DL, Levin B, Hornig M, Fiehn O, Lipkin WI. Insights into myalgic encephalomyelitis/chronic fatigue syndrome phenotypes through comprehensive metabolomics. Sci Rep. 2018 Jul 3;8(1):10056. doi: 10.1038/s41598-018-28477-9. PMID 29968805
- [Background] Nkiliza A, Parks M, Cseresznye A, Oberlin S, Evans JE, Darcey T, Aenlle K, Niedospial D, Mullan M, Crawford F, Klimas N, Abdullah L. Sex-specific plasma lipid profiles of ME/CFS patients and their association with pain, fatigue, and cognitive symptoms. J Transl Med. 2021 Aug 28;19(1):370. doi: 10.1186/s12967-021-03035-6. PMID 34454515
- [Background] Ruban A, Berkutzki T, Cooper I, Mohar B, Teichberg VI. Blood glutamate scavengers prolong the survival of rats and mice with brain-implanted gliomas. Invest New Drugs. 2012 Dec;30(6):2226-35. doi: 10.1007/s10637-012-9799-5. PMID 22392507
- [Background] Swerdlow RH, Bothwell R, Hutfles L, Burns JM, Reed GA. Tolerability and pharmacokinetics of oxaloacetate 100 mg capsules in Alzheimer's subjects. BBA Clin. 2016 Mar 10;5:120-3. doi: 10.1016/j.bbacli.2016.03.005. eCollection 2016 Jun. PMID 27051598
- [Background] Tully L, Humiston J, Cash A. Oxaloacetate reduces emotional symptoms in premenstrual syndrome (PMS): results of a placebo-controlled, cross-over clinical trial. Obstet Gynecol Sci. 2020 Mar;63(2):195-204. doi: 10.5468/ogs.2020.63.2.195. Epub 2020 Feb 25. PMID 32206660
- [Background] Vernon SD, Whistler T, Cameron B, Hickie IB, Reeves WC, Lloyd A. Preliminary evidence of mitochondrial dysfunction associated with post-infective fatigue after acute infection with Epstein Barr virus. BMC Infect Dis. 2006 Jan 31;6:15. doi: 10.1186/1471-2334-6-15. PMID 16448567
- [Background] Vidoni ED, Choi IY, Lee P, Reed G, Zhang N, Pleen J, Mahnken JD, Clutton J, Becker A, Sherry E, Bothwell R, Anderson H, Harris RA, Brooks W, Wilkins HM, Mosconi L, Burns JM, Swerdlow RH. Safety and target engagement profile of two oxaloacetate doses in Alzheimer's patients. Alzheimers Dement. 2021 Jan;17(1):7-17. doi: 10.1002/alz.12156. Epub 2020 Jul 27. PMID 32715609
- [Background] Whistler T, Taylor R, Craddock RC, Broderick G, Klimas N, Unger ER. Gene expression correlates of unexplained fatigue. Pharmacogenomics. 2006 Apr;7(3):395-405. doi: 10.2217/14622416.7.3.395. PMID 16610950
- [Background] Wilkins HM, Harris JL, Carl SM, E L, Lu J, Eva Selfridge J, Roy N, Hutfles L, Koppel S, Morris J, Burns JM, Michaelis ML, Michaelis EK, Brooks WM, Swerdlow RH. Oxaloacetate activates brain mitochondrial biogenesis, enhances the insulin pathway, reduces inflammation and stimulates neurogenesis. Hum Mol Genet. 2014 Dec 15;23(24):6528-41. doi: 10.1093/hmg/ddu371. Epub 2014 Jul 15. PMID 25027327
- [Background] Williams DS, Cash A, Hamadani L, Diemer T. Oxaloacetate supplementation increases lifespan in Caenorhabditis elegans through an AMPK/FOXO-dependent pathway. Aging Cell. 2009 Dec;8(6):765-8. doi: 10.1111/j.1474-9726.2009.00527.x. Epub 2009 Sep 30. PMID 19793063
- [Background] Yamano E, Sugimoto M, Hirayama A, Kume S, Yamato M, Jin G, Tajima S, Goda N, Iwai K, Fukuda S, Yamaguti K, Kuratsune H, Soga T, Watanabe Y, Kataoka Y. Index markers of chronic fatigue syndrome with dysfunction of TCA and urea cycles. Sci Rep. 2016 Oct 11;6:34990. doi: 10.1038/srep34990. PMID 27725700
- [Background] Yoshikawa K. Studies on the anti-diabetic effect of sodium oxaloacetate. Tohoku J Exp Med. 1968 Oct;96(2):127-41. doi: 10.1620/tjem.96.127. No abstract available. PMID 4884771
- [Derived] Cash A, Vernon SD, Rond C, Bateman L, Abbaszadeh S, Bell J, Yellman B, Kaufman DL. RESTORE ME: a RCT of oxaloacetate for improving fatigue in patients with myalgic encephalomyelitis/chronic fatigue syndrome. Front Neurol. 2024 Nov 27;15:1483876. doi: 10.3389/fneur.2024.1483876. eCollection 2024. PMID 39664752
- See also: Oxaloacetate Acid Supplementation as a Mimic of Calorie Restriction — https://benthamopen.com/contents/pdf/TOLSJ/TOLSJ-3-22.pdf